CLINICAL TRIAL: NCT06123871
Title: Expression Analysis of Urinary Exosome miR-136-5p in Type 2 Diabetic Nephropathy and Evaluation of Its Clinical Diagnostic Value
Brief Title: Expression Analysis of Urinary Exosome in Type 2 Diabetic Kidney Disease and Evaluation of Its Clinical Diagnostic Value
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yipeng Liu (Other)
Responsible Party: Sponsor-Investigator, Yipeng Liu, Clinical Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023(127)
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2 diabetes group: The group was based on the clinically confirmed diagnosis of type 2 diabetes
  Interventions: Other: Grouping based on previous laboratory results, no intervention.
- Diabetic nephropathy group: The group was based on the clinically confirmed diagnosis of type 2 diabetes.The group was based on the clinically confirmed diagnosis of type 2 diabetes.Patients were re-screened strictly according to the following admission criteria: persistent albuminuria and/or decreased eGFR,while other causes of chronic kidney disease (CKD) were excluded. When diabetes mellitus is identified as the cause of kidney damage and other primary and secondary glomerular diseases and systemic diseases are excluded, at least one of the following conditions can be diagnosed as DKD: (1) Urinary Albumin/Creatinine Ratio(UACR)≥30 mg/g or Urinary albumin excretion rate (UAER)≥30 mg/24 h, The UACR or UAER was checked again within 3 to 6 months, and 2 out of 3 times reached or exceeded the critical value; Eliminate other interfering factors such as infection; (2) eGFR< 60 ml·min-1.(1.73 m2) -1 for more than 3 months;(3) Renal biopsy was consistent with DKD pathological changes.
  Interventions: Other: Grouping based on previous laboratory results, no intervention.

INTERVENTIONS:
Other: Grouping based on previous laboratory results, no intervention. — The patients were grouped according to the results of previous inpatient tests, and no intervention measures were taken

SUMMARY:
Expression analysis of urinary exosome miR-136-5p in type 2 diabetic nephropathy and evaluation of its clinical diagnostic value

DETAILED DESCRIPTION:
1. Preliminary screening of miRNAs: Through GEO database and reading related literature, miRNAs differentially expressed in type 2 diabetes and diabetic nephropathy were selected as potential candidate biomarkers for follow-up verification.
2. Collection and treatment of clinical samples: Urine of diabetic patients was collected from the First Affiliated Hospital of Shandong First Medical University in strict accordance with the drainage standard, and the basic information of patients was registered. Meanwhile, the collected samples were divided into type 2 diabetes group and diabetic nephropathy group according to whether the urine was accompanied by UACR≥300/g. Subsequently, the collected samples were centrifuged and retained for supernatant.
3. Isolation and identification of urinary exosomes: Ultrafast centrifugation method was used to separate the treated urine samples of exosomes, and then identified by transmission electron microscopy, nanoparticle analysis and Western blot respectively.
4. Real-time PCR was used to detect the changes in urinary exosomal miRNA expression levels of the two groups of patients, and statistical analysis and correlation analysis of clinical indicators of the differentially expressed mirnas were performed.
5. Target gene prediction and enrichment pathway analysis of differentially expressed mirnas were performed to screen out pathways that might be related to the occurrence and development of DKD, and then the relevant pathways were verified by immunofluorescence, immunocoprecipitate, Western blot, Real- time PCR and other methods.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Previously diagnosed with type 2 diabetes;
3. Typical diabetic symptoms (polydipsia, polydipsia, polyuria and weight loss) plus random blood glucose ≥11.1mmol/l;
4. Fasting blood glucose ≥7.0mmol/l, fasting is defined as at least 8 hours without intake of calories;
5. Oral glucose tolerance test (OGTT) 2-hour blood glucose ≥11.1mmol/ l, using a glucose load equivalent to 75 grams of anhydrous glucose dissolved in water (venous blood was drawn in all patients;
6. With or without UACR≥300mg/g.

Exclusion Criteria:

1. Refused to enroll patients;
2. Type 1 diabetic nephropathy and other special types of diabetic nephropathy; 3.Patients with kidney stones and urinary system infection;

4.Patients with autoimmune system diseases, malignant tumors, and blood system diseases; 5.Patients with severe chronic cardiopulmonary disease, chronic liver and kidney disease; 6.Patients with severe infectious diseases; #7#Use of glucocorticoids, immunosuppressants or cytotoxic drugs.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a clinically confirmed diagnosis of type 2 diabetes during hospitalization in the Department of nephrology and Endocrinology from December 2020 to June 2022.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Preliminary screening of miRNA | 2020-2024
  Through GEO database and reading related literature, mirnas that are differentially expressed in type 2 diabetes and diabetic nephropathy were selected as potential candidate biomarkers for follow-up verification.
Clinical sample collection and processing | 2020-2024
  The urine of diabetic patients was collected from the First Affiliated Hospital of Shandong First Medical University in strict accordance with the drainage standard, and the basic information of patients was registered. Meanwhile, the collected samples were divided into type 2 diabetes group and diabetic nephropathy group according to whether the urine was accompanied by UACR≥300/g. Subsequently, the collected samples were centrifuged and retained for supernatant.
Statistical analysis and target gene prediction of misexpressed mirnas and enrichment pathway analysis | 2020-2024
  Statistical analysis and correlation analysis of clinical indicators of differenti ally expressed mirnas were performed to further evaluate their clinical diagnostic value.Subsequently, the target gen es of the mirnas differentially expressed in urinary exosomes of the two groups were analyzed by miRTarBase datab base and R software package, and the relevant pathways were screened out through KEGG enrichment pathway a analysis. Subsequently, the relevant pathways were verified by immunofluorescence, immunocoprecipitation, We estern blot, Real-time PCR and other methods.

CONTACTS AND LOCATIONS:
Overall Officials: Yipeng Liu, Study Chair — Qianfoshan Hospital
Locations (1):
- Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No